CLINICAL TRIAL: NCT00644644
Title: A Validation of the NTX Wireless Patient Monitoring System in Combination With Novel Computer Interface to Generate Proactive Medical Responses to Patient Specific Events
Brief Title: Validation of the NTX Wireless Patient Monitoring System
Acronym: TATRC
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Dan France, Associate Professor, Vanderbilt University
Other Study IDs: 061241
Record Dates: First submitted 2008-03-19; First posted 2008-03-27 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Desaturation; Bradycardia; Tachycardia; Hypertension; Hypotension
Keywords: NTX; Nihon Kohden; mobile monitoring
MeSH Terms: conditions — Bradycardia; Tachycardia; Hypertension; Hypotension | interventions — Hospital Rapid Response Team

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: monitored
  Interventions: Other: Rapid Response Team (NTX wireless monitoring system)
- 2: control

INTERVENTIONS:
Other: Rapid Response Team (NTX wireless monitoring system) — If the subject is experiencing a life threatening change in their vital signs, the Rapid Response Team will be initiated per VUMC protocol.
  Other Names: - attending nurse action per VUMC protocol
  Groups: 1

SUMMARY:
* Reduction in time to detection of Clinically Significant events
* Reduction of time to Intervention during Clinically Significant events
* Reduction in the number of admissions to Intensive Care

DETAILED DESCRIPTION:
1200 patients will have wireless monitors attached to their arm. They will be randomized to have their vital signs filtered through software that generates alerts, or software that does not generate alerts. Low and high limit alarms will be set according to published guidelines and adjusted at will by the response team. If appropriate the Vanderbilt University Medical Center Rapid Response team will be initiated per Institutional Policy

ELIGIBILITY:
Inclusion Criteria:

* Ability to give written informed consent
* Patients that are hospitalized for longer than 24 hours and are located on the 4th, 5th, or 6th floor of the Vanderbilt University Medical Center Round Wing
* Patients must be ≥18 years of age

Exclusion Criteria:

* ICU patients
* Female subjects who are pregnant
* Patients < 18 years of age
* Patients that have a contradiction for continuous Blood Pressure monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-op orthopedic and GI patients who will be admitted for a minimum of 24 hours to the Round Wing area of Vanderbilt University Medical Center.
Sampling Method: Probability Sample
Enrollment: 1303 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To determine if the NTX wireless monitoring system in combination with a novel computer interface will provide early detection of potentially life threatening changes in patient's vital signs | an interim analysis will be performed after 400 patients have been placed on the study, again after 800 have been places on the study

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J France, PhD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt University Medical Center Department of Anesthesiology — http://www.vandydreamteam.com